CLINICAL TRIAL: NCT02713633
Title: Prospective Randomized Trial of Indwelling Double-J Ureteral Stent Versus Externalized Modified-Salle Stent for Pyeloplasty
Brief Title: Indwelling Double-J Ureteral Stent Versus Externalized Modified-Salle Stent for Pyeloplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in staffing, original PI no longer at our institution.
Sponsor: Rajeev Chaudhry (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor-Investigator, Rajeev Chaudhry, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14010600
Record Dates: First submitted 2016-02-23; First posted 2016-03-21 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Ureteropelvic Junction Obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Stent (Other): we use one method, we choose were we will leave the stent and then we create a small hole in the kidney and then pull the stent through the hole and then create small hole in the abdominal fascia and then the skin, all this done under direct vision and control. So now the sent is outside the patient and connected directly to the kidney and the renal pelvis, then the distal part of the stent will be inserted across the anastomosis and before closing the renal pelvis (also under vision) toward the ureter. The external stent will be connected at the end of the procedure to a urine bag.
  Interventions: Other: internal Double-J stents; Other: External Stent
- internal Double-J stents (Other): internal stent, we use to approaches to insert it: 1- Retrograde by cystoscopy and this will take 10 minutes before starting the surgical procedure itself and we put the stent under fluoroscopy guidance and this is the commonest way we use now to put the internal stents. 2- ante grade, and this is basically inserting the stent during the surgical procedure itself from the kidney down to the ureter and this is done without fluoroscopy
  Interventions: Other: internal Double-J stents; Other: External Stent

INTERVENTIONS:
Other: internal Double-J stents — internal stent, we use to approaches to insert it: 1- Retrograde by cystoscopy and this will take 10 minutes before starting the surgical procedure itself and we put the stent under fluoroscopy guidance and this is the commonest way we use now to put the internal stents. 2- ante grade, and this is basically inserting the stent during the surgical procedure itself from the kidney down to the ureter and this is done without fluoroscopy
Other: External Stent — we use one method, we choose were we will leave the stent and then we create a small hole in the kidney and then pull the stent through the hole and then create small hole in the abdominal fascia and then the skin, all this done under direct vision and control. So now the sent is outside the patient and connected directly to the kidney and the renal pelvis, then the distal part of the stent will be inserted across the anastomosis and before closing the renal pelvis (also under vision) toward the ureter. The external stent will be connected at the end of the procedure to a urine bag.

SUMMARY:
This prospective study, Randomized Trial of Indwelling Double-J Ureteral Stent Versus Externalized Modified-Salle Stent for Pyeloplasty will consist of four steps: 1.) Enrolling subjects in the study and signing the consent form 2.) Randomly divide subjects into 2 groups, group 1 will have internal stent and group 2 will have external stent 3.) At the time of stent removal in the clinic or in the OR subjects parents/ subjects will fill a questionnaire about pain after the procedure, stent care and stent tolerance and 4) Data from the questionnaires and procedure cost will be collected and all the data will be analyzed

DETAILED DESCRIPTION:
The pyeloplasty is a surgical procedure to treat kidney obstruction due to congenital or acquired causes. Congenital like congenital stenosis in the Uretero-pelvic junction (UPJ) or due to crossing blood vessels. Acquired causes like UPJ obstruction post stone disease or renal trauma. For the congenital or the acquired causes the principle of the surgery is to remove the UPJ stenosis (the diseased segment of the ureter) and reconnect the ureter to the renal pelvis again. This procedure is known as dismembered pyeloplasty. It was described in 1940 by Anderson and since then still the gold standard procedure regardless of the approach (open, laparoscopic or robotic). One of the principles of the procedure is to 'Splint' the anastomosis, i.e put something across the anastomosis during the healing process that includes internal and external stents. Also there are surgeons even don't believe in keeping anything across the anastomosis, but they leave a nephrostomy tube only that will not cross the anastomosis. In our division at CHP, we believe that we should keep a stent across the anastomosis to help in the healing process and decrease that chance of intra-abdominal urine leak and to increase the chance of success (90-99%). So for the internal stent, we use to approaches to insert it: 1- Retrograde by cystoscopy and this will take 10 minutes before starting the surgical procedure itself and we put the stent under fluoroscopy guidance and this is the commonest way we use now to put the internal stents. 2- ante grade, and this is basically inserting the stent during the surgical procedure itself from the kidney down to the ureter and this is done without fluoroscopy. For the external stent we use one method, we choose were we will leave the stent and then we create a small hole in the kidney and then pull the stent through the hole and then create small hole in the abdominal fascia and then the skin, all this done under direct vision and control. So now the sent is outside the patient and connected directly to the kidney and the renal pelvis, then the distal part of the stent will be inserted across the anastomosis and before closing the renal pelvis (also under vision) toward the ureter. The external stent will be connected at the end of the procedure to a urine bag. The type of the procedure will not affect out choice of the type of the stent, as both stents can be inserted using the open, laparoscopic or robotic approach. No difference in the choice for antibiotics or pain medication, again because we will perform the same exact surgery (open, lap or robotic pyeloplasty) and so the same incisions. All out patients receive pre and post-operative antibiotics and this will not be different in both groups. For the alternative method, simply is choosing the first patient for example for internal stent, the second patient we will use external stent, the third patient we will use internal stent, then external , then internal..etc. We will not choose the patient according to age or sex. Of course after we tell the parents and the patient about the study and they choose not to enroll, we will use the internal stent as we usually do. Basically all the pyeloplasty surgeries (open, Lap or robotic) are done as inpatient. All the patients will spend the night in the hospital with Foley catheter and next day and after full evaluation most of the patients will be sent home. All the pyeloplasty surgeries are done under general anesthesia.

This is prospective study to compare the post-operative pain, stent tolerance, stent care and total cost of a common procedure in pediatric urology which is pyeloplasty. The patients will be randomized into 2 groups. All female subjects will undergo a standard urine pregnancy test to rule out pregnancy. The first group will be patients who will have internal Double-J stents and the second group will be patients who will have external Pippi-Salle nephron-ureteric stent. The parents and the patient will be informed at the day of the surgery about the type of stent he/she will have at the end of the surgery. In the post-operative period, the patient will stay overnight (as for all the non-study patients) and next morning his/her Foley catheter will be removed. The patient and his/her family will receive instructions about the care for external stent (if he/she has one) and receive the regular prescriptions for pain medicine and Oxybutynin (if the patient has internal stent). All patients will be given contact information to call in case they have concerns or questions about the study, the procedure itself or the stents.

Patients will be randomized to the two different post-operative stent treatments using block randomization with permuted blocks. Block randomization will help ensure that by the end of the study we have a reasonably similar number of patients in each treatment group. Given that the investigators are necessarily unmasked in this study since they are placing the stents, randomly permuted blocks will ensure that the investigators cannot identify the pattern and predict the stent the next patient will receive.

The website www.randomization.com has been used to generate a randomization schedule using block sizes of 9 and 6. This suggests an estimated 45 patients will be recruited at a single site so that across 2 institutions about 90 patients will be recruited with approximately 30 patients total per treatment group by the end of the study.

The Principal Investigator is Dr. Michael C. Ost, M.D, chief of the division of Pediatric urology with the research pediatric urology fellow Dr. Pankaj Dangel, M.D and the clinical pediatric urology fellow Dr. Moira Dwyer, M.D. All the patients' names, details of the procedures and the parents/patients questionnaires will be kept as part of medical records that is protected by the HIPPA regulations for confidentiality.

ELIGIBILITY:
Inclusion Criteria: Ureteropelvic Junction Obstruction

-

Exclusion Criteria: Pregnancy

Ages: 3 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the two different Stents | 4-6 weeks until the stent is removed
  Post-operative pain control and tolerance
Comparison of the two different Stents removal | 4-6 weeks until the stent is removed
  the ease of stent removal
Comparison of the two different Stents patient satisfaction | 4-6 weeks until the stent is removed
  Patient/parents satisfaction and cost

SECONDARY OUTCOMES:
Compare patient/parent reported tolerance | 4-6 weeks until the stent is removed
  assess the patient/parent reported outcomes for post-operative pain, tolerance
Compare patient/parent reported outcome | 4-6 weeks until the stent is removed
  ease of stent removal will be measured

OTHER OUTCOMES:
Questionnaire | 4-6 weeks until the stent is removed
  Since the validity of self-reported response is unclear at this time, data will be used to formulate future questionnaire and will be validated in set of patients. The data in the study will be presented in descriptive format for example we may find that 30% of the patients with internal stents have bladder spasms, and 40% of patients with external stents have site related pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We are sharing de-identified data with University of Chicago

REFERENCES:
- [Background] Yiee JH, Baskin LS. Use of internal stent, external transanastomotic stent or no stent during pediatric pyeloplasty: a decision tree cost-effectiveness analysis. J Urol. 2011 Feb;185(2):673-80. doi: 10.1016/j.juro.2010.09.118. Epub 2010 Dec 18. PMID 21172705
- [Result] Castagnetti M, Rigamonti W. Re: Outcome analysis and cost comparison between externalized pyeloureteral and standard stents in 470 consecutive open pyeloplasties. L. H. P. Braga, A. J. Lorenzo, W. A. Farhat, D. J. Bagli, A. E. Khoury and J. L. Pippi Salle. J Urol 2008; 180: 1693-1699. J Urol. 2009 Jul;182(1):399-400. doi: 10.1016/j.juro.2009.02.152. Epub 2009 May 20. No abstract available. PMID 19467676
- [Result] Elmalik K, Chowdhury MM, Capps SN. Ureteric stents in pyeloplasty: a help or a hindrance? J Pediatr Urol. 2008 Aug;4(4):275-9. doi: 10.1016/j.jpurol.2008.01.205. Epub 2008 Mar 7. PMID 18644529